CLINICAL TRIAL: NCT01255956
Title: Efficacy Evaluation of In-bare Metal Stent Restenosis Treatment With Rapamycin Eluting Stent or Paclitaxel Eluting Balloon Catheter. Study With Intravascular Ultrasound and Optical Coherence Tomography
Brief Title: Restenosis Treatment With Rapamycin Eluting Stent or Paclitaxel Eluting Balloon Catheter (RESTENOZA)
Acronym: ISRII
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Warsaw (Other)
Collaborators: KCRI (Other)
Responsible Party: Medical University of Warsaw, Medical University of Warsaw
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Restenoza II 4.0
Record Dates: First submitted 2010-12-06; First posted 2010-12-08 (Estimated); Last update posted 2011-01-25 (Estimated); Status verified 2011-01

CONDITIONS: In-Stent Restenosis
Keywords: restenosis; ISR; in-stent restenosis; drug eluting stent; rapamycin eluting stent; paclitaxel eluting balloon catheter

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rapamycin eluting stent (Experimental): Patients treated with rapamycin eluting stent (n=100)
  Interventions: Device: Rapamycin eluting stent implantation
- Paclitaxel eluting balloon catheter (Experimental): Patients treated with paclitaxel eluting balloon catheter (n=100)
  Interventions: Device: Paclitaxel eluting balloon catheter

INTERVENTIONS:
Device: Rapamycin eluting stent implantation — Rapamycin eluting stent implantation for in-stent restenosis treatment
  Arms: Rapamycin eluting stent
Device: Paclitaxel eluting balloon catheter — Paclitaxel eluting balloon catheter for in-stent restenosis treatment
  Arms: Paclitaxel eluting balloon catheter

SUMMARY:
The aim of the study is to compare rapamycin eluting stent and paclitaxel eluting balloon catheter in the treatment of restenosis in bare metal stent.

DETAILED DESCRIPTION:
Study aims:

* Clinical efficacy evaluation of different treatment's strategies, including periprocedural and long-term endpoints defined as: death, myocardial infarction, brain stroke, necessity of repeated revascularization
* Evaluation of intravascular ultrasound (IVUS) as an optimisation method for direct and long-term revascularization effects
* Evaluation of optical coherence tomography as an optimisation method for direct and long-term revascularization effects
* Evaluation of late lumen loss and neointimal hyperplasia in stent in long-term follow-up
* Analysis of direct and indirect medical costs of alternative treatment strategies

Study group:

200 patients with symptomatic restenosis evidenced angiographically in bare metal stent implanted in native coronary artery. Patients will be randomised to 2 therapeutic groups:

* Patients treated with rapamycin eluting stent (n=100)
* Patients treated with paclitaxel eluting balloon catheter (n=100)

ELIGIBILITY:
Inclusion Criteria:

* at least 18 years of age
* symptomatic restenosis in bare metal stent implanted in native coronary artery
* angina pectoris
* ischemia evidenced by non-invasive diagnostic tests
* angiographically evidenced in-stent restenosis > 50% assessed by quantitative coronary angiography (QCA)
* vessel diameter > 2,5 mm

Clinical exclusion criteria:

* myocardial infarction within less than past 72 hours
* heart failure with left ventricular ejection fraction (LVEF) < 30%
* chronic renal failure with significant impairment of glomerular filtration (creatinine > 2 mg/dl)
* hypersensitivity or contraindication to acetylsalicylic acid, clopidogrel, heparin, abciximab, rapamycin, paclitaxel
* hypersensitivity to contrast
* other diseases that may cause significant deterioration in long-term prognosis
* acute or chronic inflammatory diseases
* patients who are unwilling to consent for participation in the study

Angiographic exclusion criteria:

* significant stenosis in left main coronary artery (LM)
* multivessel disease qualifying for coronary artery bypass grafting (CABG)
* anatomical localization and morphology that preclude optimal percutaneous intervention intervention's (PCI) result or intravascular ultrasound (IVUS) or optical coherence tomography performance
* vessel diameter < 2,5 mm
* restenotic lesion length > 30 mm

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2010-12; Primary Completion 2012-07 (Estimated); Study Completion 2012-07 (Estimated)

PRIMARY OUTCOMES:
Incidence of repeated restenosis angiographically evidenced | at 9 months
Neointimal volume assessed by intravascular ultrasound (IVUS) | at 9 months
Late lumen loss and neointimal volume assessed by optical coherence tomography (OCT) | at 9 months

SECONDARY OUTCOMES:
Incidence of repeated target lesion revascularization (TLR) | at 9 months
Incidence of repeated target vessel revascularization (TVR) | at 9 months
Incidence of death | at 9 months
Incidence of myocardial infarction | at 9 months
Incidence of brain stroke | at 9 months
Incidence of in-stent thrombosis | at 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Jacek Legutko, MD, PhD, Principal Investigator — II Department of Cardiology Medical College Jagiellonian University University Hospital in Krakow
Locations (4):
- Poland (4):
  - Instytut Kardiologii w Warszawie-Aninie, Warsaw, Alpejska 42
  - Katedra i Klinika Kardiologii Warszawskiego Uniwersytetu Medycznego, Warsaw, Banacha 1a
  - Klinika Kardiologii z Kliniką Kardiochirurgii Uniwersyteckiego Szpitala Klinicznego w Lodzi, Lodz, Kniaziewicza 1/5
  - II Department of Cardiology Medical College Jagiellonian University University Hospital in Krakow, Krakow, Kopernika 17